CLINICAL TRIAL: NCT02236871
Title: FAMILY (FAmily MILk Product Two-Year) Dose-response Study to Enhance Bone Health
Brief Title: Family Milk Product Two-year Dose-response Study to Enhance Bone Health
Acronym: FAMILY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University (Other)
Collaborators: Dairy Farmers of Canada (Other)
Responsible Party: Principal Investigator, Hope Weiler, Associate Professor, McGill University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HW-14-03
Record Dates: First submitted 2014-09-04; First posted 2014-09-11 (Estimated); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Healthy
Keywords: Adolescents; Dairy; Bone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control (No Intervention): Maintain current milk and milk product intakes.
- 2 servings (Active Comparator): Participants will be asked to consume 1 milk (250 ml) plus a yogurt (100-175 g) or cheese (up to 50 g) to reach an average of 2 servings of milk or milk products/d.
  Interventions: Behavioral: 2 servings
- 4 servings (Active Comparator): Participants will be asked to consume recommended servings of milk or milk products/d for their age, so they will receive 1 milk (250 ml), a yogurt (175 g) and cheese (50 g) or more. This would provide ≥ 3 servings/d.
  Interventions: Behavioral: 4 servings

INTERVENTIONS:
Behavioral: 2 servings — Participants will receive motivational counseling to help the improve milk and milk product intakes to 2 servings per day.
  Arms: 2 servings
Behavioral: 4 servings — Participants will receive motivational counseling to help them increase their milk and milk product intake to 4 servings per day.
  Arms: 4 servings

SUMMARY:
The final stages in the development of peak bone mass (PBM) reside in late adolescence or early adulthood and are critical in the achievement of bone health. Optimization of PBM and maintenance of bone mineral density (BMD) are the best population health strategies in the primary prevention of osteoporosis. Diet and activity are key lifestyle factors in the primary prevention of osteoporosis as recognized in Canada's Food and Activity Guides. Dietary Reference Intakes are evidence-based regarding nutrition and bone health with a focus on calcium and vitamin D; yet the Food Guide and health behaviors are reliant on actual foods. The number of recommended servings of milk and alternatives varies by age with average intakes estimated to be below targets for all Canadians > 9 y of age. This is especially concerning during development of PBM. Therefore, the global objective is to generate high-level evidence that dietary intervention with milk and milk products will enhance PBM in young men and women and maintenance of BMD in their parents.

The primary objective is to demonstrate in healthy young men and women (14-18.9 y at baseline) with habitually low usual milk and milk product intakes that intervention with greater milk and milk product consumption improves lumbar spine BMD in a dose-response manner over 2 y (while accounting for body size, physical activity, demographics and age). Healthy young men and women will be recruited and screened for usual intake of milk and milk products. Those with low intakes < 2 servings of milk or milk products will be randomized (stratified by sex and age) to 1 of 3 groups for the RCT (n=10090/group): maintain usual low intakes (<1 serving), improved intakes (average of 2 servings/d) or recommended intakes (≥3 servings/d) of milk and milk products. A manualized motivational interviewing framework will be used for the interventions. Those meeting recommendations at screening will form a longitudinal cohort for 2 y. Key measurements include baseline and yearly assessment of BMD at multiple sites plus interim assessment of general health, anthropometry, dietary intakes, physical activity and biomarkers of calcium homeostasis; and in the young adults bone metabolism.

DETAILED DESCRIPTION:
Rationale:

The final stages in development of peak bone mass (PBM) take place in late adolescence or early adulthood and are vital for attaining optimal bone health. The variation in bone mineral density (BMD) at the time of PBM is similar with aging, suggesting that the benefits of efforts to enhance BMD early will later be realized with aging. Therefore, optimization of PBM and maintenance of BMD are thus the best population health strategies in the primary prevention of osteoporosis and reduction in risk of fracture.

Osteoporosis is a bone disease that results in low bone mass and reduced bone tissue, thereby, increasing bone fragility. The World Health Organization (WHO) defines osteoporosis as a BMD value of 2.5 SD or more below a reference population specific PBM and is associated with an elevated risk of fracture. Diet and activity are key lifestyle factors in the primary prevention of osteoporosis. The number of recommended servings of milk and alternatives varies by age with actual intakes estimated to be below targets for all Canadians 9 y of age and older. For example, young men and women, aged 15 to 18.9 years, should consume 3 to 4 servings/day of milk and alternatives according to Canada's Food Guide, however, in reality, adherence to food guide recommendations is not the norm for Canadians with intakes as low as 1.36 servings in males and 1.24 servings in females on average.

If Canadians are to realize the benefits of meeting Canada's Food Guide recommended servings for the Milk and Alternates Food Group, at least in terms of meeting nutrient intake recommendations if not bone health outcomes, behavior change will be necessary. There is some evidence that increasing milk and/or milk products is a proven approach to achieving calcium intake with benefits to bone health. From a professional counselling perspective, motivational interviewing techniques have been useful in stimulating and sustaining behavior change given its success in triggering changes in a number of health behaviors.

Besides counseling, research suggests that the family environment or social support system predict ability to make behavior change. Healthy physical activity and nutrition are reliant upon parental behaviors, beliefs and perceptions and may also include practical parental support for modeling healthy food intake or accessibility to healthy food at home. Therefore, studying the role of parents in increasing their children's dairy intake will be of an added-value to our study.

Research Center:

All of the objectives will be exclusively tested at one research centre, the Mary Emily Clinical Nutrition Research Unit of McGill University. This unit is administratively linked to the School of Dietetics and Human Nutrition for which Dr. Weiler is the Director.

Population:

Healthy young men and women (n=270) 14 to 18.9 y of age from the Greater Montreal Area residing with their parent(s); one 14 to 18.9 y per household will be included.

Design:

Parallel randomized controlled dose-response trial using milk and milk products as the main source of calcium in 14 to 18.9 y young men and women (n=270) from the Greater Montreal area for 2 years of study.

Methodology of Research:

Males and females (14-18.9 y) with habitual milk and milk products intake < 2 servings/d will be randomized (random numbers tables) to one of the three groups below; stratified based on sex and age to ensure balanced groups. All will be asked to consume a milk serving and milk products, examples are below. For this study milk can be skim, 1%, 2% or whole, cheeses are not processed (e.g. select regular cheddar, mozzarella) and yogurts may be of variable milk fat content.

DETAILS OF MEASUREMENTS

Demographics:

Upon written consent, a demographics survey will be completed with parents that include age and education of parents, family income range and employment. Parents will be asked to self-identify ethnicity for themselves and the participating child to facilitate understanding of the relationships among culture, skin pigmentation and baseline vitamin D status.

Anthropometry:

In the fasting state, weight and height will be measured using standard clothing and a calibrated balance-beam scale and a wall-mounted stadiometer to calculate BMI. Waist circumference will be measured according to Health Canada guidelines. Body composition will be measured every 6 mo using BIA as a rapid assessment.

Health Measures:

General health history and adverse events over the previous 6 mo will be documented by survey. At baseline, 1y and 2y, all participants will have their heart rate and blood pressure measured by a registered nurse. A short-form Profile of Mood States (POMS) will be taken baseline and yearly.

Activity:

For our study, the International Physical Activity Questionnaire (iPAQ) will be completed at baseline and every 6 mo to determine physical activity level; participants may also be asked to wear accelerometers (tri-axial ActiGraph GT3X (ActiGraph LLC, Fort Walton Beach, FL) to further capture activity over 2 weekdays and 2 weekend days prior to each visit as a more objective measure of activity.

Dietary Intake Survey:

A FFQ (modified Harvard) for use in English or French (25) and tested in adults will be used to capture past intakes (1 y) at baseline, 12 and 24 mo. Dietary intakes will also be captured using 24-h recalls at baseline, 1, 3 and 6 mo and at 6 mo intervals thereafter. Telephone calls will be every 3 months with both the child and the parent on the line to improve compliance to group.

Exposure to UVB:

To help explain vitamin D and for skin type, exposure to UVB (i.e. endogenous synthesis of vitamin D) will be assessed at each visit using changes in skin pigmentation at constitutive (inner upper arm) and facultative (forehead, mid-forearm and lower leg) sites using a spectrophotometer. Travel and UVB exposure including clothing habits (eg, short sleeves, shorts hats etc.) and use of sun blocks (UVB level and frequency of use etc) will be surveyed as well. Measurements performed on the unexposed skin of the inner upper arm have higher correlation to the Melanin Index than measurements performed on the exposed forehead according to standard guidelines.

Bone Mass Assessment:

The minimum detectable change in areal BMD (aBMD) using DXA is ~1% for all types of scans. In order to confidently examine changes in BMD following interventions in young adults, study duration is 2 y. Whole body, LS vertebrae 1 to 4 (AP and lateral), left hip (total and FN) and forearm (non-dominant) will be measured using a Hologic 4500A fan-beam clinical densitometer at baseline, 1 and 2 y. For this test, RCT participants will wear standardized clothing (cotton pants and T-shirts). DXA is rapid, taking a total of 5-7 minutes x-ray time, and the low radiation (<10 uSV) will not exceed limits for x-ray exposure. Values will be compared to the Hologic normative databases and thus expressed as BMC and BMD along with Z-scores where applicable (from the National Health and Nutrition Examination Survey [NHANES] reference database) and from CaMos data. Quality control data will be monitored and maintained using a proprietary LS bone phantom (Hologic). To complement, tibia and forearm BMD will be measured at baseline, 1 and 2 y as well using the peripheral quantitative computed tomography technique (pQCT). Unlike most other common techniques for measuring BMD, a pQCT scan is able to measure volumetric bone mineral density and the geometry of the bone whereas DXA is only able to provide the areal bone mineral density. For this measurement we will examine sites ranging from 4 to 66% from the distal radius and tibia of the non-dominant side; the 4% site will provide for a trabecular rich region and the 66% will provide a cortical bone assessment, we will also examine the 14% and 38% sites of the tibia.

Sample Procurement:

All blood samples (2x 8-10 ml tubes) will be collected at the Mary Emily Clinical Nutrition Research Unit on the Macdonald Campus of McGill University between 0700 and 1000 h in the fasted state (minimum 8 h) and separated into plasma (~ 4 ml) and serum (~4 ml) fractions and immediately measured for analytes or stored at -80 oC until analysis; analytes susceptible to degradation on freeze thaw (OC) will be measured only on samples thawed once

Details of Biochemistry:

Vitamin D (25(OH)D), osteocalcin (OC) and PTH concentration will be measured the same day (or batched monthly) using a Liaison autoanalyzer (DiaSorin): Total Vitamin D (sensitivity: 4 ng/ml); bioactive PTH kit (sensitivity <4 pg/ml) and OC (sensitivity 0.3 ng/mL) kits. In batches, manual ELISA will be used for CTX. Ionized calcium will be measured on-site using a radiometer blood gas tube within 4 h of collection; this will also provide us with hemoglobin and hematocrit concentrations. Total serum plus urinary calcium and creatinine and lipid assessments including serum HDL, LDL and total cholesterol (LDL) and triacylglycerols will be measured through the MUHC clinical laboratory fee for service system.

ELIGIBILITY:
Inclusion Criteria:

* 14 to 18.9 y of age at onset of the intervention
* reside with their parents
* consume < 1 serving/d of milk and milk products
* > 2 y post-menarche
* non smoker
* not routinely taking prescribed oral medication including oral/dermal
* healthy body mass index (BMI) defined as ± 1SD of 50% percentile WHO curves
* normal bone mass for age/sex
* adequate vitamin D status (>30 nmol/L 25(OH)D)
* no anemia
* receptive to stop any nutritional supplements 2 weeks prior to and during the study.

Exclusion Criteria:

* Any known chronic disease with exception of mild asthma (<500 µg budesonide) that does not affect BMD Z-scores
* Anaemic (defined as Hg <13.5 g/dL in males and <12.0 g/dL in females for their age group).
* Known allergies or aversions to milk and milk products
* Anticipating becoming pregnant or a moving distant from Montreal or from family home in the next 2 y.
* Have preference for non-dairy alternatives
* consume ≥2 alcoholic beverages/day

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 94 (Actual)
Dates: Start 2014-05; Primary Completion 2019-12-20 (Actual); Study Completion 2019-12-20 (Actual)

PRIMARY OUTCOMES:
Change in lumbar spine BMD (g/cm2) at 2 years. | up to 2 years
  To examine in healthy young men and women (14-18.9 y at baseline) with habitually low usual milk and milk product intakes (<1 serving/d) whether intervention with greater milk and milk product consumption improves lumbar spine (LS) BMD at 2 years in a dose-response manner.

SECONDARY OUTCOMES:
Change in calcium homeostasis at 2 years. | up to 2 years
  To explore if calcium homeostasis is altered by milk intake.
Change in whole body BMD (g/cm2) at 2 years | up to 2 years
  Examine the difference in whole body BMD (g/cm2) at 2 years
Change in total hip BMD (g/cm2) at 2 years. | up to 2 years
Change in distal forearm BMD (g/cm2) at 2 years. | up to 2 years
Change in femoral neck BMD (g/cm2) at 2 years. | up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Hope A Weiler, PhD, Principal Investigator — McGill University
Locations (1):
- Mary Emily Clinical Nutrition Research Unit, Sainte-Anne-de-Bellevue, Quebec, Canada

REFERENCES:
- See also: Research site website — http://www.mcgill.ca/mecnru